CLINICAL TRIAL: NCT05993273
Title: Pain Control After VATS Anatomical Pulmonary Resections: Randomized Comparison Between Cryoanalgesia, Erector Spinae Plane Block and Epidural Catheter
Brief Title: Pain Control After VATS Anatomical Pulmonary Resections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Giovanni Maria Comacchio, Thoracic Surgeon, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5697/AO/23
Record Dates: First submitted 2023-07-25; First posted 2023-08-15 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer; Pain, Postoperative; Thoracic Neoplasms
Keywords: thoracoscopic surgery; post-operative pain; epidural anesthesia; ESP block; cryoanalgesia; lobectomy
MeSH Terms: conditions — Lung Neoplasms; Pain, Postoperative; Thoracic Neoplasms | interventions — Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Epidural (Experimental): In patients randomized to this Arm, before the induction of general anesthesia, the epidural catheter is placed in the intervertebral space (T4-T5, T5-6 or T6-T7) and used intra and post-operatively for administration of local anesthetics.
  Interventions: Procedure: Epidural
- ESP block (Experimental): In patients randomized to this Arm, after induction of general anesthesia the Erector spinae plane (ESP) block is performed with a catheter introduced and left in place for continuous postoperative infusion of local anesthetics.
  Interventions: Procedure: ESP block
- Cryoanalgesia (Experimental): In patients randomized to this Arm, after induction of general anesthesia and single lung ventilation the first thoracoscopic surgical access is performed. A cryoanesthesia device with a dedicated atraumatic angled-tip cryoprobe is inserted through the thoracoscopic access and the active tip of the probe is positioned in contact with the intercostal nerves from T3 to T8.
  Interventions: Procedure: Cryoanalgesia

INTERVENTIONS:
Procedure: Epidural — The epidural catheter is placed while the patient is awake, before the induction of general anesthesia. The intervertebral spaces used for catheter insertion are alternatively T4-T5, T5-6 or T6-T7. After locating the epidural space through the technique of the loss of resistance, a catheter is introduced for about 5 cm and left in place for the administration of drugs into the epidural space. Once the correct functioning of the epidural catheter has been verified with a negative test for cerebrospinal fluid aspiration and a negative bolus test for the onset of signs and symptoms from intrathecal infusion, the catheter is used intraoperatively for administration of local anesthetics in refracted boluses (Lidocaine and Ropivacaine ) at anesthetic dosage and postoperatively for continuous infusion of Ropivacaine 0.15% at 5 mL/h.
  Arms: Epidural
Procedure: ESP block — Erector spinae plane (ESP) block is performed after induction of general anesthesia, with the patient in a lateral decubitus position. With the aid of the ultrasound guide with linear probe, the transverse process of T5 ipsilateral to the site of the operation is identified. With the in-plane technique, the lower fascia of the ESP muscle is hydrodissected through the administration of Ropivacaine 0.5% 3 mg/Kg lean body weight. Subsequently, a catheter is introduced and left in place for continuous postoperative infusion of Ropivacaine 0.2% at 12 mL/h.
  Arms: ESP block
Procedure: Cryoanalgesia — Cryoanalgesia is performed after the induction of general anesthesia, single lung ventilation and after performing the first thoracoscopic surgical access. A cryoanesthesia device with a dedicated atraumatic angled-tip cryoprobe is inserted through the thoracoscopic access. The active tip of the probe is positioned in contact with the intercostal nerves from T3 to T8 and kept resting for 4 ½ minutes on each nerve at a temperature of -70°C, under direct thoracoscopic vision, generating an interruption of the sensory functions.
  Arms: Cryoanalgesia

SUMMARY:
In patients undergoing minimally invasive thoracoscopic surgery (video-assisted thoracoscopic surgery, or VATS), moderate to severe post-operative pain may often be experienced. The presence of pain negatively affects the perceived quality of care and can predispose to complications, as the development of chronic pain.

In order to prevent post-operative pain, different multimodal pain treatment protocols are applied, consisting in combinations of local-regional anesthesiological techniques and intravenous medications.

Regional anesthesia is considered essential to prevent pain in the immediate post-operative period. However, to date, there is no agreement regarding which is the most effective regional anesthesiological technique; therefore, the choice is usually based on the Anesthetist's preferences.

The aim of this study is to compare three regional anesthesiological techniques (cryoanalgesia, epidural anesthesia, and erector spinae muscle plane block) routinely used during thoracoscopic lung surgery.

DETAILED DESCRIPTION:
In patients undergoing minimally invasive thoracoscopic surgery (video-assisted thoracoscopic surgery, or VATS), moderate to severe post-operative pain may often be experienced. The presence of pain negatively affects the perceived quality of care and can predispose to complications, as the development of chronic pain.

In order to prevent post-operative pain, different multimodal pain treatment protocols are applied, consisting in combinations of local-regional anesthesiological techniques and intravenous medications.

Regional anesthesia is considered essential to prevent pain in the immediate post-operative period. However, to date, there is no agreement regarding which is the most effective regional anesthesiological technique; therefore, the choice is usually based on the Anesthetist's preferences.

The aim of this study is to compare three regional anesthesiological techniques (cryoanalgesia, epidural anesthesia, and erector spinae muscle plane block) routinely used during thoracoscopic lung surgery.

All patients undergoing anatomical pulmonary resections (lobectomy or segmentectomy) through a thoracoscopic (VATS) approach, and who present the inclusion/exclusion characteristics, will be considered.

The day of surgery, patients are randomized 1:1:1 to receive 3 different pain control techniques: epidural catheter, ESP block or cryoanalgesia.

A standard pain management protocol will be applied to all patient after surgery.

Primary Outcome Measure is the perceived post-operative pain 24 hours after surgery in the 3 groups, evaluated through numeric pain rating scale (NPRS). Other outcome measures are the post-operative pain trend and the patients' total amount of opioid use in the postoperative period (expressed as Morphine milligram equivalents).

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing VATS anatomic pulmonary resection (lobectomy or segmentectomy) for benign or malignant disease

Exclusion Criteria:

* Refusal or inability to give informed consent to the study protocol
* Age < 18 years
* Pregnancy
* Allergies or contraindications to any of the treatments considered in the experimental design
* Pre-operative use of pain medication for chronic pain or neuropathic pain
* History of previous major chest surgery
* American Society of Anesthesiologists (ASA) class > 3
* Need for intensive care unit stay in the post-operative period
* Patients undergoing anatomical pulmonary resections different than lobectomy or segmentectomy (bi-lobectomy or pneumonectomy).
* Patients undergoing bronchial and/or vascular resections and reconstructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 24 hours after surgery
  Perceived post-operative pain 24 hours after surgery through Numeric Pain Rating Scale (NPRS, value from 0 to 10, o=no pain, 10=worst pain ever)

SECONDARY OUTCOMES:
Post-operative pain trend | 1,6,12 and 48 hours after surgery
  Perceived post-operative pain 1,6,12 and 48 hours after surgery through Numeric Pain Rating Scale (NPRS, value from 0 to 10, o=no pain, 10=worst pain ever)
Rescue Analgesia | 48 hours after surgery
  patients' total amount of opioid use in the postoperative period (expressed as Morphine milligram equivalents)

CONTACTS AND LOCATIONS:
Overall Officials: MARCO MAMMANA, MD, PhD, Principal Investigator — PADUA UNIVERSITY HOSPITAL
Locations (1):
- Thoracic Surgery Unit, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005
- [Background] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Sepsas E, Misthos P, Anagnostopulu M, Toparlaki O, Voyagis G, Kakaris S. The role of intercostal cryoanalgesia in post-thoracotomy analgesia. Interact Cardiovasc Thorac Surg. 2013 Jun;16(6):814-8. doi: 10.1093/icvts/ivs516. Epub 2013 Feb 19. PMID 23424242
- [Background] Ju H, Feng Y, Yang BX, Wang J. Comparison of epidural analgesia and intercostal nerve cryoanalgesia for post-thoracotomy pain control. Eur J Pain. 2008 Apr;12(3):378-84. doi: 10.1016/j.ejpain.2007.07.011. Epub 2007 Sep 17. PMID 17870625
- [Background] Torre M, Mameli L, Bonfiglio R, Guerriero V, Derosas L, Palomba L, Disma N. A New Device for Thoracoscopic Cryoanalgesia in Pectus Excavatum Repair: Preliminary Single Center Experience. Front Pediatr. 2021 Jan 18;8:614097. doi: 10.3389/fped.2020.614097. eCollection 2020. PMID 33585365
- [Background] Lin J, Liao Y, Gong C, Yu L, Gao F, Yu J, Chen J, Chen X, Zheng T, Zheng X. Regional Analgesia in Video-Assisted Thoracic Surgery: A Bayesian Network Meta-Analysis. Front Med (Lausanne). 2022 Apr 6;9:842332. doi: 10.3389/fmed.2022.842332. eCollection 2022. PMID 35463038
- [Background] Fiorelli S, Leopizzi G, Menna C, Teodonio L, Ibrahim M, Rendina EA, Ricci A, De Blasi RA, Rocco M, Massullo D. Ultrasound-Guided Erector Spinae Plane Block Versus Intercostal Nerve Block for Post-Minithoracotomy Acute Pain Management: A Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2020 Sep;34(9):2421-2429. doi: 10.1053/j.jvca.2020.01.026. Epub 2020 Jan 21. PMID 32144056
- [Background] Taketa Y, Irisawa Y, Fujitani T. Comparison of ultrasound-guided erector spinae plane block and thoracic paravertebral block for postoperative analgesia after video-assisted thoracic surgery: a randomized controlled non-inferiority clinical trial. Reg Anesth Pain Med. 2019 Nov 8:rapm-2019-100827. doi: 10.1136/rapm-2019-100827. Online ahead of print. PMID 31704789